CLINICAL TRIAL: NCT03876067
Title: The Cardioprotective Effects of Adding Ozone To Cardioplegic Solution in Adult Cardiac Surgery
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Israa mohamed lotfallah, assistant lecture assiut university hospital principle investigator, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: AssuitUlotfallah
Record Dates: First submitted 2019-03-10; First posted 2019-03-15 (Actual); Last update posted 2019-03-19 (Actual); Status verified 2019-03

CONDITIONS: Ischemic Heart Disease
MeSH Terms: conditions — Myocardial Ischemia | interventions — Ozone; Cardioplegic Solutions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ozone Group (Experimental): in which Ozone will be added to cold blood cardioplegia
  Interventions: Drug: Ozone
- Control Group (Placebo Comparator): : in which in which only cold blood cardioplegia
  Interventions: Drug: Cardioplegic Solutions

INTERVENTIONS:
Drug: Ozone — Our procedures for O3T application in CBP surgery conform to international guidelines of the ''Madrid Declaration on Ozone Therapy'' 32 . M-O3T will be carried out as follows:
  50mL of blood drawn by vacuum from the patient central catheter into a sterile blood transfusion bag in which 10 mL of 3.8% Na citrate solution (Galenica Senese Industries, Siena, Italy) as an anticoagulant will be previously added so that the blood/citrate volume ratio was 9:1. After blood withdrawal, the bag will momentarily disconnected leaving the venous access open by a saline infusion 33 . A corresponding volume (50 mL) of gas was immediately added with an O3 concentration of 20-50 micrograms/mL gas. Ozone was produced by Medozon compact generator (Herrmann Apparatebau GmbH, Germany).
  At this point, the hyper-oxygenated ozonated blood will be mixed with the cold cardioplegia (Thomsons cardioplegia) this amount of ozonated blood will be added to each 500 ml of cardioplegic solution
  Arms: Ozone Group
Drug: Cardioplegic Solutions — in which in which only cold blood cardioplegia
  Arms: Control Group

SUMMARY:
forty patients with age ranged between 40-70 years undergoing elective coronary artery bypass graft surgery with cardiopulmonary bypass will be included, they will divided into two groups.

Ozone Group: in which Ozone will be added to cold blood cardioplegia. Control Group: in which in which only cold blood cardioplegia

Primary outcome:

Pattern of recovery of myocardium after declamping of Aorta

1. Time of cardiac rhythm return after declamping.
2. type of cardiac rhythm after declamping and rate of DC use.

Secondary outcome:

A-cardiac parameters

* Post operative inotropic score
* Incidence of post operative cardiac dysrhythmias
* postoperative ejection fraction (EF)
* Postoperative parameters of myocardial ischaemia
* a- Troponin levels
* b-Pro BNP
* • Histopathology of myocardial sample for detection of myocyte cellular edema as a marker of ischemic changes.

B-non cardiac parameters:

1. inflammatory markers 1. CRP 2. L\N 3. P\N
2. ICU stay
3. hospital stay
4. morbidity and mortality

DETAILED DESCRIPTION:
Ozone Administration Protocol

Our procedures for O3T application in CBP surgery conform to international guidelines of the ''Madrid Declaration on Ozone Therapy'' 32 . M-O3T will be carried out as follows:

50mL of blood drawn by vacuum from the patient central catheter into a sterile blood transfusion bag in which 10 mL of 3.8% Na citrate solution (Galenica Senese Industries, Siena, Italy) as an anticoagulant will be previously added so that the blood/citrate volume ratio was 9:1. After blood withdrawal, the bag will momentarily disconnected leaving the venous access open by a saline infusion 33 . A corresponding volume (50 mL) of gas was immediately added with an O3 concentration of 20-50 micrograms/mL gas. Ozone was produced by Medozon compact generator (Herrmann Apparatebau GmbH, Germany).

The gas is immediately and continuously mixed with the blood in the bag for at least 5 min and with gentle rotating movement to avoid foaming. Due to the blood viscosity, the gas mixture does not instantaneously come into contact with the whole blood mass, thus this mixing time is necessary. During these 5 min of mixing, the ozone totally reacted with both the potent antioxidants of plasma and the unsaturated lipids bound to albumin, generating asmall amount of hydrogen peroxide and alkenals. These two messengers were responsible for eliciting crucial biochemical reactions on both erythrocytes and within cells. At this point, the hyper-oxygenated ozonated blood will be mixed with the cold cardioplegia (Thomsons cardioplegia) this amount of ozonated blood will be added to each 500 ml of cardioplegic solution

Exclusion Criteria:

The patient will be excluded from the study if he has any of the following:

* left ventricular ejection fraction< 40%
* diabetic or other metabolic disorders,
* use of left ventricular assist devices,
* Renal failure or on hemodialysis
* Hepatic dysfunction
* Hypothyroidism
* implanted pacemaker

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective CABG surgery

Exclusion Criteria:

* • left ventricular ejection fraction< 40%

  * diabetic or other metabolic disorders,
  * use of left ventricular assist devices,
  * Renal failure or on hemodialysis
  * Hepatic dysfunction
  * Hypothyroidism
  * implanted pacemaker

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-04-01 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Time of cardiac rhythm | one hour
  Time of cardiac rhythm return after declamping.
type of cardiac rhythm | one hour
  type of cardiac rhythm after declamping and rate of DC use

SECONDARY OUTCOMES:
Post operative inotropic score | two weeks
  Post operative inotropic score
post operativecardiac dysrhythmias | two weeks
  Incidence of post operativecardiac dysrhythmias
postoperative ejection fraction (EF) | one month
  postoperative ejection fraction (EF)
Postoperative parameters of myocardial ischaemia | two weeks
  Troponin levels
ICU stay | two weeks
  ICU stay
mortality | two weeks
  mortality